CLINICAL TRIAL: NCT02641938
Title: Effect of Intraoperative Dexmedetomidine on Development of Acute Kidney Injury Following Cytoreduction and Hyperthermic Intraperitoneal Chemotherapy: a Double-blind Randomized Clinical Trial
Brief Title: Effect of Intraoperative Dexmedetomidine on Development of Acute Kidney Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-young Kim, Associate Professor, Yonsei University Medical College, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3-2015-0262
Record Dates: First submitted 2015-12-20; First posted 2015-12-30 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): 1ug/kg IV loading over 20 minutes followed by 0.5ug/kg/hr IV infusion after induction of anesthesia until the completion of the surgery
  Interventions: Drug: Dexmedetomidine
- Normal Saline (Placebo Comparator): IV loading and infusion of same volume of normal saline after induction of anesthesia until the completion of the surgery
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine group :1ug/kg IV loading over 20 minutes followed by 0.5ug/kg/hr IV infusion after induction of anesthesia until the completion of the surgery
  Arms: Dexmedetomidine
Drug: Normal Saline — Control group :IV loading and infusion of same volume of normal saline after induction of anesthesia until the completion of the surgery
  Arms: Normal Saline

SUMMARY:
To investigate the renal protective effect of dexmedetomidine in patients undergoing cytoreduction and hyperthermic intraperitoneal chemotherapy

DETAILED DESCRIPTION:
A cytoreductive surgery and hyperthermic intraperitoneal chemotherapy may lead to the renal hypoperfusion, systemic inflammatory response, and oxidative stress. Dexmedetomidine has been known to protect the kidney against inflammation and oxidative stress in diverse clinical settings. It may also enhance a renal perfusion by inhibition of renal sympathoexcitation. We hypothesized administration of dexmedetomidine might protect the kidney in patients undergoing cytoreduction and hyperthermic intraperitoneal chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant tumor with peritoneal metastasis
* Scheduled for elective cytoreduction and hyperthermic intraperitoneal chemotherapy

Exclusion Criteria:

* Preoperative chronic kidney disease stage ≥4 defined by KDOQI ( eGFR < 30 mL/min/1.73m2)
* Congestive heart failure
* Atrioventricular block > 1st degree
* Bradycardia < 45 beat per minute
* History of myocardial infarction within 3 months
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change of Creatinine clearance from baseline | Postoperative day 1,2,3,4,5,6,7
  Assessment of the creatinine clearance which reflects kidney function during postoperative 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Kim, MD, Principal Investigator — Yonsei University Medical College Gangnam Severance Hospital
Locations (1):
- GangnamSH, Seoul, South Korea

REFERENCES:
- [Derived] Song Y, Kim DH, Kwon TD, Han DW, Baik SH, Jung HH, Kim JY. Effect of intraoperative dexmedetomidine on renal function after cytoreductive surgery and hyperthermic intraperitoneal chemotherapy: a randomized, placebo-controlled trial. Int J Hyperthermia. 2019;36(1):1-8. doi: 10.1080/02656736.2018.1526416. Epub 2018 Oct 25. PMID 30354794